CLINICAL TRIAL: NCT00471809
Title: Childhood Asthma Research and Education (CARE) Network Trial - Montelukast or Azithromycin for Reduction of Inhaled Corticosteroids in Childhood Asthma (MARS)
Acronym: MARS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The CARE Network DSMB recommended to the NHLBI that the MARS trial be terminated, based on a futility analysis with 55 randomized children.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 447; 5U10HL064313 (NIH); 5U10HL064288 (NIH); 5U10HL064305 (NIH); 5U10HL064295 (NIH); 5U10HL064287 (NIH); 5U10HL064307 (NIH)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2012-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Salmeterol Xinafoate; Azithromycin; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Budesonide + Salmeterol + Azithromycin
Drug: Budesonide + Salmeterol + Montelukast
Drug: Budesonide + Salmeterol + Placebo

SUMMARY:
The MARS trial is a randomized, double-blind, parallel group study that compares the capacity of azithromycin or montelukast to placebo as effective adjunctive therapy that allows reduction of inhaled corticosteroids in children ages 6 to 17 years with moderate to severe persistent asthma. The primary null hypothesis is that in children with moderate-to-severe persistent asthma, a macrolide antibiotic (azithromycin) or a leukotriene receptor antagonist (montelukast) will provide a steroid-sparing effect when compared to placebo as the dose of inhaled corticosteroid is reduced. This will be tested following achievement of control of symptoms with moderate to high-dose inhaled corticosteroid in combination with a long-acting bronchodilator agonist. Use of these doses for the inhaled corticosteroid will be based on NHLBI step-up guidelines to achieve asthma control.

DETAILED DESCRIPTION:
The MARS trial is a randomized, double-blind, parallel group study that compares the capacity of azithromycin or montelukast to placebo as effective adjunctive therapy that allows reduction of inhaled corticosteroids in children ages 6 to 17 years with moderate-to-severe persistent asthma. The primary null hypothesis is that in children with moderate-to-severe persistent asthma, a macrolide antibiotic (Mac - azithromycin) or a leukotriene receptor antagonist (LTRA - montelukast) will provide a steroid-sparing effect when compared to placebo as the dose of inhaled corticosteroids (ICS - budesonide) is reduced. This will be tested following achievement of control of symptoms with moderate to high-dose ICS in combination with a long-acting bronchodilator agonist (LABA - salmeterol). Use of these doses for the inhaled corticosteroid will be based on NHLBI step-up guidelines to achieve asthma control. Inadequate asthma control is defined as either:

1. chronic poor control: a) symptoms, or albuterol use for symptoms or low peak flow, or peak flow less than 80% baseline on greater than 3 days per week on average, or b) nocturnal awakenings for asthma symptoms requiring albuterol 2 or more nights over 2 weeks of observation, or c) FEV1 less than 80% of the best pre-randomization value on 2 consecutive visits 1-4 days apart, or
2. an asthma exacerbation as determined by need for systemic corticosteroids

Treatment in the run-in period will be determined by the child's status at the first visit. At enrollment (V0) all patients will be given budesonide as the ICS and salmeterol as the LABA. Children will be treated with salmeterol BID and a dose of ICS based on chronic medication use with stepping-down based on time and symptoms until criteria for inadequate control as indication for stepping-up the dose of ICS. When inadequate control is documented (V1), a four-day course of prednisone will be administered and the dose of ICS (still administered with salmeterol BID) will be doubled to establish control. The children will be followed with monthly clinic visits and interim phone calls, emphasizing use of daily diary to document symptoms and doses of albuterol required. Reestablishment of control during a 2-week interval will prompt randomization. If control is not yet established by the first increase in ICS dose during the stabilization period, the dose can be doubled along with a second prednisone course until a maximum of budesonide of 1600 mcg/day is attained. The daily dose of budesonide at randomization will be a minimum of 800 mcg to allow for a maximum of 4-fold reduction of dose, and a maximum of 1600 mcg to allow for patient safety considering side effects of high dose ICS.

When clinical control is achieved by the increased dose of ICS, a child will then be randomized (V2) to one of the three treatment arms, (1) placebo (one placebo tablet and one or two placebo capsules), (2) azithromycin (one placebo tablet and one or two capsules containing azithromycin with the dose based on weight), or (3) montelukast (one tablet containing montelukast with the dose based on age as indicated in the package insert and one or two placebo capsule). Children will be followed for an additional six weeks on the dose of ICS that achieved control ("1X") + salmeterol BID with the study medication (V3). They will then undergo three 6-week periods of ICS reduction (V4, V5, V6), first to ¾ of the control dose ("0.75X"), then ½ of the control dose ("0.5X") and then ¼ of the control dose ("0.25X"), each using salmeterol BID as concomitant medication. The ICS dosing and salmeterol will be open-label. Criteria for treatment failure and discharge from the study will be an established set of criteria that indicate reappearance of inadequate control of asthma or an exacerbation of asthma.

At the end of the double-blind administration of oral study medication (V6), patients not discharged from the study because of having met one of the criteria for inadequate control of asthma will have their study medication discontinued, with subjects continuing to take placebo capsules in addition to ¼ ICS plus salmeterol. They will then be followed for an additional 6-week single-blind wash-out period with an interim contact by phone at 3 weeks to determine the course of asthma control to determine the persistence of effect off of the study medication (V7).

The procedures to be performed at V0 are informed consent, pregnancy test, complete physical exam, spirometry, and bronchodilator response. The procedures to be performed at V1 are spirometry, complete blood count, blood IgE and eosinophils, brief physical exam, EKG, and genotyping. The following procedures will be performed at each of V2 through V7: brief physical exam, spirometry, forced oscillometry, exhaled nitric oxide, asthma control questionnaire, asthma-specific quality-of-life questionnaire, and sinusitis questionnaire. In addition, allergy skin testing will be performed at V2, pregnancy tests at V2 through V6, methacholine challenge at V2 and V3, and polymerase chain reaction for atypical organisms and macrolide antibiotic resistance (nasal wash) at V2, V5, and V7.

Finally, children will maintain daily diary records of morning and evening symptoms, peak expiratory flow rates, and rescue medication use.

ELIGIBILITY:
Inclusion Criteria:

At Enrollment (V0):

* Age 6-17 years at time of enrollment. A goal of 33% minority and 40% female subjects will be incorporated in recruitment
* Weighs at least 25 kg
* Asthma diagnosed by a physician and present for at least one year prior to study entry
* Moderate to severe persistent asthma:

  1. Patients will be identified in the following general categories. The general principle is that patients will be uncontrolled on a relatively low dose of ICS that can be stepped-up, or controlled on a moderate or high dose of ICS that can be stepped-down.

     i) On low dose ICS with or without salmeterol and uncontrolled. This patient will be treated with budesonide and salmeterol to determine eligibility criteria. If the addition of salmeterol results in control of symptoms, the patient would be excluded from MARS. If control was not established on low dose budesonide and salmeterol, the dose of budesonide would be increased and entry criteria evaluated based on the algorithm in Figure 1.

     ii) On a dose of ICS equivalent to budesonide at 400 mcg per day with or without any other medication and uncontrolled. This patient will be treated with budesonide and salmeterol to determine eligibility criteria.

     iii) On a dose of ICS equivalent to budesonide at 800 mcg per day with or without any other medication and controlled.

     iv) On a dose of ICS equivalent to budesonide at 1600 mcg per day with or without any other medication and uncontrolled but not requiring prednisone acutely. These patients will be followed to see if they become well controlled with increased adherence or more careful monitoring of symptoms.
  2. Examples are given for Advair as this drug is a commonly used form of ICS and LABA:

     i) Patients on Advair 100/50 bid and inadequately controlled ii) Patients on Advair 250/50 bid and inadequately controlled iii) Patients on Advair 250/50 bid and well controlled for greater than 3 months and being considered for stepping-down to Advair 100/50 iv) Patients well controlled on Advair 100/50 bid + either montelukast or theophylline for greater than 3 months and being considered for stepping-down to Advair 100/50 bid alone v) Patients on Advair 500/50 bid and well controlled for greater than 3 months and being considered for stepping-down to Advair 250/50 vi) Patients well controlled on Advair 250/50 bid + either montelukast or theophylline for greater than 3 months and being considered for stepping-down to Advair 250/50 bid alone
  3. Patients on an equivalent of budesonide 400 mcg, 800 mcg, or 1600 mcg per day with no symptoms, but with an FEV1 less than 80% predicted, will be enrolled as uncontrolled and observed closely for symptoms or low peak flows for 2 weeks. The rationale for enrolling these patients and observing them as "uncontrolled" is that patients with an FEV1 below the range of normal may be having symptoms and/or low peak flows that will become apparent under close observation after appropriate education. Note that a percent predicted value for FEV1 will be used only at the enrollment visit, with criteria for control and inadequate control during both run-in and during the double-blind portions of the study using the highest FEV1 value obtained during run-in for decisions prior to randomization and the FEV1 at randomization for decisions subsequent to that visit.
* FEV1 at least 80% predicted if there is going to be step-down at enrollment or at least 50% predicted if already suboptimally controlled historically and to be observed for 2 weeks to define baseline symptoms. FEV1 measurements will be obtained pre-bronchodilator.
* Demonstrate a bronchodilator response with an improvement in FEV1 of at least 12% or airway responsiveness to methacholine with a PC20 less than 12.5 mg/ml.

  1. Bronchodilator responsiveness testing will be done at Visit 0 (Enrollment) in all patients using 4 puffs albuterol.
  2. Methacholine challenge will be done at Visit 1 (Step-up) in patients who did not respond to bronchodilator at Visit 0. Patients with a FEV1 less than 70% predicted or an upper respiratory infection at the time of Visit 1 will have a second bronchodilator challenge rather than a methacholine.
* Varicella immunization complete (unless the subject has already had clinical varicella). If the subject needs varicella vaccine, this will be arranged with the primary care physician and must be received prior randomization
* Willingness to provide informed consent by the child's parent or guardian
* Nonsmoker in the past year; in addition, no use of smokeless tobacco products in the year prior to study entry

Exclusion Criteria:

At Enrollment (V0):

* More than four courses of systemic corticosteroids for asthma during the 12 months prior to study entry
* More than one hospitalization for wheezing illnesses within the 12 months prior to study entry
* Current treatment with antibiotics for diagnosed sinus disease
* History of severe sinusitis requiring sinus surgery within the past 12 months
* Use of maintenance oral or systemic antibiotics for treatment of an ongoing condition
* Use of macrolide antibiotics within the 6 weeks prior to study entry
* Requirement for prednisone therapy for concurrent illness, e.g., RA, SLE, IBD
* Asthma exacerbation requiring systemic corticosteroids within 4 weeks of study entry
* Contraindication for use of macrolide or LTRA
* Presence of lung disease other than asthma, such as cystic fibrosis and bronchopulmonary dysplasia. Evaluation during the screening process will assure that an adequate evaluation of other lung diseases has been performed
* Presence of other significant medical illnesses (cardiac, liver, gastrointestinal, endocrine, any seizure disorder except febrile seizure in infancy) that would place the study subject at increased risk of participating in the study
* Use of digoxin, ergotamine or dihydroergotamine, triazolam, carbamazepine, cyclosporine, hexobarbital, and phenytoin, and similar classes of medication will be specifically excluded
* Use of omalizumab within one year of study entry
* Gastroesophageal reflux symptoms not controlled by standard medical therapy
* Immunodeficiency disorders
* History of respiratory failure requiring mechanical ventilation for asthma within 5 years
* History of hypoxic seizure due to asthma
* Inability of the child to ingest the study drug
* Participation presently or in the past month in another investigational drug trial
* Evidence that the family may be unreliable or nonadherent, or may move from the clinical center area before trial completion
* Pregnant or breastfeeding
* Receiving hyposensitization therapy other than an established maintenance (continuous for 3 months duration or longer) regimen

At Randomization (V2):

* Still uncontrolled on step-up dosing of 1600 mcg budesonide + salmeterol BID
* Abnormal liver enzyme laboratory test results
* Abnormal QTc interval or evidence of a rhythm abnormality
* Failure to complete diary cards at expected levels (at least 75% of days) during the observation period
* Failure to adhere with oral medication use at least 80% during run-in
* Need for oral corticosteroids for a reason other than Step Up during run-in period

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210
Dates: Start 2006-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time to inadequate asthma control | Measured at Visit 7

SECONDARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | Measured at Visit 7
Mean peak flow variability | Measured at Visit 7
Asthma symptom scores | Measured at Visit 7
Overall asthma control | Measured at Visit 7
Quality of life | Measured at Visit 7
Sinusitis questionnaires | Measured at Visit 7
Exhaled nitric oxide (eNO) | Measured at Visit 7
Rescue medication use | Measured at Visit 7

CONTACTS AND LOCATIONS:
Overall Officials: Vernon M. Chinchilli, PhD, Principal Investigator — Penn State College of Medicine; Stanley J. Szefler, MD, PhD, Principal Investigator — National Jewish Health; Robert F. Lemanske, Jr., MD, Principal Investigator — University of Wisconsin, Madison; Robert S. Zeiger, MD, PhD, Principal Investigator — Kaiser Permanente Medical Center; Robert C. Strunk, MD, Principal Investigator — Washington University School of Medicine; Fernando D. Martinez, MD, Principal Investigator — University of Arizona College of Medicine; Lynn M. Taussig, MD, Study Chair — University of Denver
Locations (6):
- United States (6):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Los Angeles, Kaiser Permanente Allergy Department, Los Angeles, California
  - Kaiser Permanente Medical Center, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin - Madison, Madison, Wisconsin

REFERENCES:
- [Result] Strunk RC, Bacharier LB, Phillips BR, Szefler SJ, Zeiger RS, Chinchilli VM, Martinez FD, Lemanske RF Jr, Taussig LM, Mauger DT, Morgan WJ, Sorkness CA, Paul IM, Guilbert T, Krawiec M, Covar R, Larsen G; CARE Network. Azithromycin or montelukast as inhaled corticosteroid-sparing agents in moderate-to-severe childhood asthma study. J Allergy Clin Immunol. 2008 Dec;122(6):1138-1144.e4. doi: 10.1016/j.jaci.2008.09.028. Epub 2008 Oct 25. PMID 18951618
- See also: Childhood Asthma Research and Education (CARE) Network — http://www.asthma-carenet.org